CLINICAL TRIAL: NCT03742830
Title: Awake Intubation in Difficult Airway- a Prospective Observational Study
Brief Title: Awake Intubation V-MAC VS
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01454
Record Dates: First submitted 2018-11-09; First posted 2018-11-15 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Intubation;Difficult

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: C-MAC VS — C-MAC VS, Karl Storz AG, 78532 Tuttlingen, Germany It has a flexible tip and a distal angular offset, in which the camera and light sources are integrated. It can be aligned (up to 60°) to the patient's anatomical structures to facilitate intubation.

SUMMARY:
Nowadays, the gold standard for difficult airway management is awake intubation with a flexible fiberscope. Alternatively, when the flexible fiberscope is unable to facilitate tracheal intubation, rigid stylets may be used. One newly developed rigid video stylet also features a flexible tip (C-MAC VS, Karl Storz AG, 78532 Tuttlingen, Germany). The distal angular offset of the C-MAC VS, in which the camera and light sources are integrated, can be aligned (up to 60°) to the patient's anatomical structures to facilitate intubation.

Although awake intubation is less comfortable for the patient and more time consuming, there are several reasons why this is often performed. The investigators plan a prospective observational with 36 participants using the C-MAC VS on adult patients with indication for awake oral intubation.

To ease the placement of the tube (intubation), the investigators will use local anesthesia of the mucosa in the mouth, pharynx and larynx.

The main purpose of the study is to prove the feasibility of successful awake intubation with the C-MAC VS in adult patients. If the new device proves reliable in facilitating awake oral, future patients benefit from an additional tool that allows fast and safe intubation in difficult airway situations.

DETAILED DESCRIPTION:
In the majority of cases, airway management is uncomplicated and a straightforward procedure. Nevertheless, in rare cases complications are associated with notably high rates of serious consequences.

Therefore, assured and reliable intubation is fundamental to safe anesthetic practice.

Various approaches were introduced by the medical device industry to optimize intubation procedure. Nowadays, the gold standard for difficult airway management is awake intubation with a flexible fiberscope. Alternatively, when the flexible fiberscope is unable to facilitate tracheal intubation, rigid stylets may be used. One newly developed rigid video stylet also features a flexible tip (C-MAC VS, Karl Storz AG, 78532 Tuttlingen, Germany). The C-MAC VS is an advancement of the rigid "Bonfils" stylet (Karl Storz, Karl Storz AG, 78532 Tuttlingen, Germany). The distal angular offset of the C-MAC VS, in which the camera and light source are integrated, can be aligned (up to 60°) to the patient's anatomical structures to facilitate intubation.

Although awake intubation is less comfortable for the patient and more time consuming, there are several reasons why this is often performed.

In this research project, the investigators plan a prospective observational study using the C-MAC VS on adult patients with indication for awake oral intubation. Spontaneous ventilation will be maintained until confirmation of tracheal intubation.To ease the placement of the tube (intubation), the investigators will use local anesthesia of the mucosa in the mouth, pharynx and larynx.

The study physician will intubate the trachea of the patient using the C-MAC VS. Another person of the study team will record the primary and secondary outcomes on the Case Report Form.

After intubation, the anesthetist evaluates the intubation. Participants will be followed up for procedure related complications after the intubation and on the 1st post-anesthesia day to evaluate patient intubation comfort (VAS 1: very easy to 10: very hard).

The main purpose of the study is to prove the feasibility of successful awake intubation with the C-MAC VS in adult patients. If the new device proves reliable in facilitating awake oral, future patients benefit from an additional tool that allows fast and safe intubation in difficult airway situations.

ELIGIBILITY:
Inclusion Criteria:

* indication for awake oral intubation
* elective surgery
* age 18-80
* written Informed Consent
* knowledge of the German language enough to understand the Informed Consent

Exclusion Criteria:

* emergency patients
* uncooperative patients
* ASA (= Physical Status Classification System) V
* study equipment and personal not available

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing general anaesthesia for an elective prodcedure at the University Hospital of Bern will be screened using the Anästhesie Informations System (AIS). If a patient meets our inclusion/exclusion criteria, the investigators will visit him personally and confirm, that all criteria are met. Then, written informed consent will be obtained and the study can begin.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Intubation success | 120 seconds
  The intubation success rate at first attempt in less than 120 seconds

SECONDARY OUTCOMES:
Airway- and intubation data | Device passes patients lips until the device is completely removed out of the tracheal tube and the first end tidal CO2 is shown (the entire process should not pass 120 seconds)
  Interim times of airway management (intubation start, first view of vocal cords, device out of the tube - first end tidal CO2)
Duration of the airway management | Device passes patients lips until the device is completely removed out of the tracheal tube and the first end tidal CO2 is shown (the entire process should not pass 120 seconds)
  The period of time that is needed for the airway management and the respiratory security
Patient's comfort during intubation | On the 1st post-procedure day
  The investigators will evaluate their comfort during intubation on the 1st post-procedure day on a VAS (visual analogue pain scale) 1-10 (1: very easy, 10: very hard).
Total number of intubation attempts | The first time the device passes patients lips until the respiratory is secured so the device is completely removed out of the tracheal tube and the first end tidal CO2 is shown.
  The total number that is needed to secure the airway with intubation
Patients demographic data such as weight | During the process of screening, up to 24 hours before the study session starts
  The weight of each patient will be presented in kilograms
Patients demographic data such as size | During the process of screening, up to 24 hours before the study session starts
  The size of each patient will be presented in meter/centimeter
Patients demographic data such as gender | During the process of screening, up to 24 hours before the study session starts
  The gender (female or male) will be presented
Patients demographic data such as BMI | During the process of screening, up to 24 hours before the study session starts
  Weight and Height will be combined to report BMI in kg/m2
Patients vital parameter such as blood pressure | Device passes patients lips until the device is completely removed out of the tracheal tube and the first end tidal CO2 is shown (the entire process should not pass 120 seconds)
  The investigators will use the standard non-invasive monitoring of the University Hospital to measure the blood pressure (in millimeters of mercury)
Patients vital parameter such as heart rate | Device passes patients lips until the device is completely removed out of the tracheal tube and the first end tidal CO2 is shown (the entire process should not pass 120 seconds)
  The investigators will use the standard non-invasive monitoring of the University Hospital to measure the heart rate (beats per minute)
Patients vital parameter such as the arterial oxygen saturation | Device passes patients lips until the device is completely removed out of the tracheal tube and the first end tidal CO2 is shown (the entire process should not pass 120 seconds)
  The investigators will use the standard non-invasive monitoring of the University Hospital to measure the arterial oxygen saturation (SaO2 in percent)
The anesthetist rates the patients airway | Device passes patients lips until the device is completely removed out of the tracheal tube and the first end tidal CO2 is shown (the entire process should not pass 120 seconds)
  The anesthetist rates the POGO (Percentage of Glottis Opening), the quality of the vision device and the intubation difficulty on a VAS (visual analogue pain scale) 1-10 (1: very easy, 10: very hard).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, Prof.Dr.med., Principal Investigator — University Hospital of Bern, Bern, Switzerland
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Background] Ovassapian A. The flexible bronchoscope. A tool for anesthesiologists. Clin Chest Med. 2001 Jun;22(2):281-99. doi: 10.1016/s0272-5231(05)70043-5. PMID 11444112
- [Background] Falcetta S, Pecora L, Orsetti G, Gentili P, Rossi A, Gabbanelli V, Adrario E, Donati A, Pelaia P. The Bonfils fiberscope: a clinical evaluation of its learning curve and efficacy in difficult airway management. Minerva Anestesiol. 2012 Feb;78(2):176-84. Epub 2011 Nov 18. PMID 22095109